CLINICAL TRIAL: NCT02911857
Title: An Extension Study of CACZ885N2301 (NCT02059291), Multi-center, Open Label Study of Canakinumab in Japanese Patients With Periodic Fever Syndromes (Tumor Necrosis Factor Receptor Associated Periodic Syndrome (TRAPS), Hyper Immunoglobulin D Syndrome ((Also Known as Mevalonate Kinase Deficiency) (HIDS/MKD), or Colchicine Resistant/Intolerant Familial Mediterranean Fever (crFMF))
Brief Title: An Extention Study of Safety of Canakinumab in Japanese Patients With Periodic Fever Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885N2301E2
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: Periodic Fevers Syndrome
Keywords: Canakinumab,; interleukin-1; Periodic Fevers Syndrome; TRAPS; HIDS; crFMF; auto-inflammatory diseases; extension study
MeSH Terms: interventions — canakinumab; secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canakinumab (ACZ885) (Experimental): Participants continued the study drug based on the final dose and regimen administered at the end of the CACZ885N2301 study. All participants received 1 or 2 ACZ885 subcutaneous injections every 4 or 8 weeks.
  Interventions: Biological: Canakinumab (AIN457)

INTERVENTIONS:
Biological: Canakinumab (AIN457) — Canakinumab solution for subcutaneous injection in vial which contained 150mg/mL canakinumab in 1 mL solution

SUMMARY:
The primary objective of this study was to evaluate safety and tolerability of ACZ885 in this extension study. This extension study offered the opportunity for participants who completed Epoch 4 of the preceding CACZ885N2301 (NCT02059291) study to continue to be treated with ACZ885 until approval in Japan of the drug in Periodic Fever Syndromes or until development of ACZ885 in Periodic Fever Syndromes was suspended.

ELIGIBILITY:
Inclusion Criteria:

* Completed Epoch 4 of the CACZ885N2301 study in Japan before the approval of canakinumab in Japan
* Written informed consent. Parent or legal guardian's written informed consent and child's assent, if appropriate, are required before any assessment is performed for patients < 20 years of age

Exclusion Criteria:

* Any conditions or significant medical problems in which the investigator judges the patient should not enter this extension study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with Tumor Necrosis Factor Receptor Associated Periodic Syndrome (TRAPS), Hyper Immunoglobulin D Syndrome (also known as mevalonate kinase deficiency (HIDS/MKD), or colchicine resistant/intolerant Familial Mediterranean Fever (crFMF) received study drug based on the final dose regimen received in CACZ885N2301 (NCT02059291).
Groups:
- TRAPS; HIDS/MKD; cfFMF: Participants continued the study drug based on the final dose and regimen administered at the end of the CACZ885N2301 study. All participants received 1 or 2 ACZ885 subcutaneous injections every 4 or 8 weeks.
Period: Overall Study
Arm/Group | TRAPS | HIDS/MKD | cfFMF
Started | 2 | 1 | 1
Completed | 2 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRAPS | HIDS/MKD | cfFMF | Total
Number analyzed (Participants) | 2 | 1 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.0 (2.83) | 14 (NA) — There is only 1 participant in the HIDS/MKD group. Therefore, standard deviation does not apply. | 20 (NA) — There is only 1 participant in the cfFMF group. Therefore, standard deviation does not apply. | 18.5 (3.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events, Serious Adverse Events and Deaths
Description: Participants were monitored for safety throughout the study.
Time Frame: Participants were followed for the duration until approval, an expected average of 3 months.
Population: Safety set: The safety set included all participants who were treated in this extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | TRAPS | HIDS/MKD | cfFMF
Number analyzed (Participants) | 2 | 1 | 1
Participants
  Non-serious adverse events | 1 | 1 | 0
  Serious adverse events | 0 | 0 | 0
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- TRAPS: TRAPS
- HIDS: HIDS
Arm/Group | TRAPS | HIDS | cfFMF
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRAPS (N=2) | HIDS (N=1) | cfFMF (N=1)
NASOPHARYNGITIS (Infections and infestations) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT02911857/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02911857/SAP_001.pdf